CLINICAL TRIAL: NCT07051811
Title: A Prospective, Multicenter, Blinded, Randomized Controlled Clinical Trial Evaluating the Safety and Efficacy of a Single-Use Intravascular Ultrasound Ablation Catheter and Ultrasound Ablation System in the Treatment of Primary Hypertension
Brief Title: To Evaluate the Safety and Efficacy of a Single-Use IVUS Ablation for Primary Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPCTP-2021-004(CT)
Record Dates: First submitted 2025-06-24; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-02

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal denervation (RDN) Group (Experimental): Receive standardized treatment with a minimum of two drugs and renal denervation treatments (RDN)
  Interventions: Procedure: Intravascular Ultrasound Ablation Therapy
- Control Group (Sham Comparator): Receive standardized treatment with a minimum of two drugs and renal artery angiography only
  Interventions: Procedure: Renal Artery Angiography

INTERVENTIONS:
Procedure: Intravascular Ultrasound Ablation Therapy — The single-use intravascular ultrasound ablation catheter is used in conjunction with the ultrasound ablation device to remove renal sympathetic nerves.
  Standardized medication regimen.
  Arms: Renal denervation (RDN) Group
Procedure: Renal Artery Angiography — Only undergo renal artery angiography. Standardized medication regimen.
  Arms: Control Group

SUMMARY:
This is a prospective, multicenter, blinded, randomized controlled clinical trial designed to evaluate the safety and efficacy of a single-use intravascular ultrasound ablation catheter and ultrasound ablation system in the treatment of primary hypertension.

DETAILED DESCRIPTION:
This trial adopts a prospective, multicenter, randomized controlled design to validate the safety and efficacy of a single-use intravascular ultrasound ablation catheter and ultrasound ablation system in the treatment of primary hypertension. Subjects who signed the informed consent form will enter the screening phase and undergo a run-in period for 4-week of standardized medication regimen. Specifically, their current antihypertensive treatment will be uniformly replaced with a combination of an angiotensin II receptor blocker (ARB) and calcium channel blocker (CCB) (Valsartan/Amlodipine 80:5 mg) or a triple combination of ARB/CCB (Valsartan/Amlodipine 80:5 mg) plus a diuretic (Hydrochlorothiazide 12.5mg) . If the subject's office systolic blood pressure (SBP) ≥180 mmHg or diastolic blood pressure (DBP) ≥110 mmHg during the run-in period, the investigator may adjust the medication and restart a run-in period of ≥28 days. Blood pressure will be re-evaluated, and subjects failed to meet the inclusion criteria after adjustment will be excluded.

Subjects meeting the inclusion criteria and not violating exclusion criteria will be randomized in a 2:1 ratio to either the treatment group or the control group. The treatment group will undergo intravascular ultrasound ablation therapy, while the control group will only undergo renal artery angiography. Both groups will maintain the standardized medication regimen for 6 months post-procedure (if a subject's office SBP exceeds 180 mmHg or drops below 110 mmHg in three consecutive measurements spaced 1 hour apart, the investigator may adjust the medication and record their blood pressure before the adjustment).

The primary efficacy endpoint is the change in 24-hour average ambulatory systolic blood pressure at 6 months post-procedure. Results will be analyzed using a superiority testing hypothesis to demonstrate that the treatment group achieves significantly greater reduction in 24-hour mean ambulatory systolic blood pressure compared to the control group at 6-month follow-up. During follow-up, office blood pressure, 24-hour ambulatory blood pressure, medication usage, safety events, and adverse events will be recorded for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years and ≤75 years, regardless of gender.
2. Documented history of primary hypertension.
3. Stable use of at least two antihypertensive medications for a minimum of 4 consecutive weeks prior to randomization, specifically requiring a combination of an angiotensin II receptor blocker (ARB) and a calcium channel blocker (CCB) or a triple combination of ARB/CCB plus a diuretic agent . After at least 4 consecutive weeks of screening, blood pressure must meet the following criteria:

   1. Office systolic blood pressure (SBP) ≥150 mmHg and <180 mmHg;
   2. Office diastolic blood pressure (DBP) ≥90 mmHg;
   3. 24-hour ambulatory systolic blood pressure ≥135 mmHg and <170 mmHg.
4. Patients who can understand the purpose of the trial, voluntarily participate and sign the informed consent form, and are willing to comply with clinical follow-up.

Exclusion Criteria:

1. Unsuitable Renal Artery Anatomy for Treatment

   1. Main renal artery diameter <4 mm or length <20 mm.
   2. Accessory renal artery diameter ≥ 2 mm and <4 mm.
   3. Renal artery stenosis >50% in the main renal artery.
   4. Renal artery aneurysm, fibromuscular dysplasia, or severe calcification.
   5. Presence of a renal artery stent.
   6. Single kidney.
2. Estimated Glomerular Filtration Rate (eGFR) <45 mL/min/1.73 m².
3. Diagnosis of Type 1 Diabetes Mellitus.
4. Orthostatic Hypotension.
5. Recent Vascular Events:Acute myocardial infarction, unstable angina, syncope, or cerebrovascular accident within 3 months prior to signing the informed consent form.
6. Suspected Secondary Hypertension.
7. Respiratory Support:a) Requirement for long-term oxygen support or mechanical ventilation (excluding nocturnal respiratory support for sleep apnea).
8. Prior Renal Artery Denervation Procedure.
9. Life Expectancy <1 Year.
10. Pregnancy, Lactation, or Plans to Become Pregnant Within 6 Months (for Females); Males Planning to Conceive Within 6 Months.
11. Current Participation in Another Clinical Trial Without Completion of the Primary Endpoint.
12. Allergy to Contrast Agents.
13. Other Reasons Deemed by the Investigator to Make the Subject Unsuitable for Participation (e.g., Poor Compliance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour average ambulatory systolic blood pressure (SBP) [at 6 months post-procedure] | From baseline to 6 months

SECONDARY OUTCOMES:
Change in Daytime/Nighttime Average Ambulatory Systolic Blood Pressure (SBP) | 1 Month, 2 Months, and 6 Months Post-Procedure
Change in 24-Hour/Daytime/Nighttime Average Ambulatory Diastolic Blood Pressure (DBP) | 1 Month, 2 Months, and 6 Months Post-Procedure
Change in 24-Hour Average Ambulatory Systolic Blood Pressure (SBP) | 1 Month and 2 Months Post-Procedure
Change in Office Systolic Blood Pressure | 1 Month, 2 Months, and 6 Months Post-Procedure
Change in Office Diastolic Blood Pressure | 1 Month, 2 Months, and 6 Months Post-Procedure
Achievement Rate of Target Office Systolic Blood Pressure | 1 Month, 2 Months, and 6 Months Post-Procedure
Composite Index of Antihypertensive Medication Use | 1 Month, 2 Months, and 6 Months Post-Procedure
Proportion of Subjects with ≥5 mmHg Reduction in 24-Hour Average Ambulatory Systolic Blood Pressure | 6 Months Post-Procedure

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Beijing Anzhen hospital , Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Shenzhen University General Hospital, Shenzhen, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Inner Mongolia People's Hospital, Hohhot, Neimenggu
  - Yinchuan First People's Hospital, Yinchuan, Ningxia
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No